CLINICAL TRIAL: NCT05392244
Title: The Profiles of Peripheral Blood Lymphocyte Subsets and Risk Factor of Infection in Children With Primary Nephrotic Syndrome
Brief Title: Characteristics of Peripheral Blood Lymphocyte Subsets in Children With PNS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-076
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Lymphocyte Disorder; Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- active group: Active PNS was defined as a serum albumin concentration of <2.5 g/dL and a urinary protein excretion of >40 mg/m2 per hour with high cholesterol levels.
- partial remission group: Partial remission PNS was defined as symptoms between active group and complete remission group.
- complete remission group: PNS in remission was defined as no proteinuria using the colorimetric qualitative test and a urinary protein/creatinine ratio of <0.2 on a random urine sample.

SUMMARY:
The etiology and precipitating factors of PNS remain unclear. Dysfunction of immunologic function is a classic theory of the pathogenesis of PNS. This study was aimed at investigating the characteristics of peripheral blood lymphocyte subsets and exploring its value of predicting infection in children with primary nephrotic syndrome (PNS).

DETAILED DESCRIPTION:
As a common type of nephrosis in children, primary nephrotic syndrome (PNS) is a clinical syndrome characterized by a heavy proteinuria, hypoalbuminemia, edema, and hyperlipidemia, caused by increased plasma protein permeability of the glomerular filtration membrane. To date, the etiology and precipitating factors of PNS remain unclear. Dysfunction of immunologic function is a classic theory of the pathogenesis of PNS, especially dysfunction of lymphocytes and lymphocyte subsets.

Lymphocyte subsets level can reflect human cellular immune function, which performs different biological functions, and coordinate with each other to maintain the body's immune function homeostasis. At present, many studies have shown that abnormal cellular immune function is closely related to the pathogenesis of PNS in children. Compared with children with PNS with mild proteinuria, CD8+ T cells were significantly increased in children with large proteinuria, and CD4+ T cells were reduced compared with healthy children and children with stable phase. NK cells are also considered to be an indicator that can assess the prognosis of children with PNS. Abnormal number or function of Regulatory T cells (Treg) may be involved in the occurrence of PNS proteinuria, and the urine protein level of the rat model can be relieved by the increase of Treg cells. Although studies have found abnormalities in the lymphocyte subsets of children with PNS, these conclusions are not consistent, indicating that the relationship between cellular immunity and the pathogenesis of children with PNS remains to be studied.

Children with PNS are susceptible to various of infections. After the application of glucocorticoids, children with PNS are more susceptible to infection, even if the infection is not serious, which can lead to recurrence of PNS or affect the curative efficacy of treatment. Studies have found that corticosteroid therapy affects the distribution of lymphocyte subsets in children with PNS, and changes in the level of CD4+ T cells are related to the occurrence and severity of infection in children with NS. The above studies all indicate that lymphocyte subsets analysis has important research significance in the occurrence and prevention of infections in children with PNS.

In this study, we observed the profiles of peripheral blood lymphocyte subsets in healthy children and children with PNS, and explored the risk factor of infection in children with PNS.

ELIGIBILITY:
Inclusion Criteria:

* age <18 years old
* first PNS episode or PNS in remission
* no history of corticosteroid or immunosuppressor use in the four weeks prior to disease occurrence

Exclusion Criteria:

* Subjects with infantile (or congenital) nephrotic syndrome (NS), secondary NS, glomerulonephritis, or systemic disease were excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From September, 2019 to April, 2021, a total of 89 children who were admitted in the Nanfang Hospital Affiliated to Southern Medical University and met the Evidence-based Guidelines for the Diagnosis and Treatment of Children's Hormone Sensitivity, Relapsed/Dependent Nephrotic Syndrome (2016), were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05-30 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
peripheral blood lymphocyte subsets | 2019.9-2020.12
  The percentage and absolute counts of lymphocyte subsets were conducted with a BD Canto Ⅱ flow cytometry (FCM)
biochemical indicators | 2019.9-2020.12
  biochemical indicators which were related to PNS, including 24-hour urine protein (UTP), serum albumin (ALB), serum total cholesterol (CHOL) and serum creatinine (Scr) were collected

IPD SHARING:
Plan to Share IPD: Undecided